CLINICAL TRIAL: NCT05545176
Title: The Validation and Development of Termination-of-Resuscitation (TOR) Rules in Patients Following Out-of-Hospital Cardiac Arrest (OHCA) in Asia Countries
Brief Title: The Validation and Development of Termination-of-Resuscitation (TOR) Rules in OHCA Patients in Asia Countries
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 202206030RINC
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-07

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out-Of-Hospital Cardiac Arrest; OHCA
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- out of hospital cardiac arrest patients in Asia countries
  Interventions: Other: termination of resuscitation rules

INTERVENTIONS:
Other: termination of resuscitation rules — Use retrospective data to analyze the accuracy termination of resuscitation rules and further develope a termination of resuscitation rule.

SUMMARY:
Objectives/Hypotheses

1. Prehospital termination-of-resuscitation (TOR) rules were developed in North American and European sites. Whether they remained valid in different geographic, ethnic, and cultural background areas is still under debate.
2. Differences in characteristics of out-of-hospital cardiac arrests (OHCAs) and configurations of emergency medical service (EMS) between the Western and Asian countries, including relatively lower rate of presenting shockable rhythm (i.e. ventricular fibrillation / ventricular tachycardia; VF/VT), lower rates of bystander CPR, less advanced life support (ALS) implementation, and less public access defibrillators, might create potential threats to the prediction accuracy of TOR rules.
3. We aim to conduct a study to validate the performance of ever published TOR rules in Asian OHCA population, including non-traumatic, traumatic, and pediatric OHCA patients. Furthermore, assess the possible variables that may impact the performance of TOR rules.
4. We also aim to develop new TOR rules based on PAROS registry for Asia population, focusing on non-traumatic, traumatic, and pediatric OHCA patients, respectively.

ELIGIBILITY:
Inclusion Criteria:

* out of hospital cardiac arrest (OHCA) patients

Exclusion Criteria:

* age <18 years
* non-EMS transport to the emergency department
* obvious signs of death (e.g. decapitation, rigor mortis, lividity, and decapitation) or having do-not-resuscitate (DNR) orders
* missing data despite meeting the inclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population included adults, OHCA patients since1 January 2007, identified from the PAROS registry. The PAROS data encompass 13 countries. The exclusion criteria include: (1) age <18 years, (2) non-EMS transport to the emergency department, (3) obvious signs of death (e.g. decapitation, rigor mortis, lividity, and decapitation) or having do-not-resuscitate (DNR) orders, and (4) missing data despite meeting the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 140000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2032-06-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
survival to hospital discharge | survival to 30-day hospitalisation
  survival to 30-day hospitalisation

SECONDARY OUTCOMES:
Cerebral Performance Categories Scale (CPC) | CPC within 30-day hospitalisation
  CPC Scale 1~5, minimum value: 1; maximum value:5; lower score means greater outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hsien Hsu, MPH, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 30 years
Access Criteria: PAROS study members